CLINICAL TRIAL: NCT06713915
Title: Diagnostic Performance of Contrast-Enhanced Mammography in Suspicious Breast Lesions
Brief Title: Diagnostic Performance of Contrast-Enhanced Mammography
Status: Not yet recruiting | Type: Observational
Sponsor: ZHOU Yidong (Other)
Responsible Party: Sponsor-Investigator, ZHOU Yidong, Breast Surgery Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: PUMCH-breast-CEM
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Mammography
Keywords: breast cancer; breast ultrasound; contrast enhanced mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- prospective cohort: Women with suspected breast abnormalities in prospective cohort will be prospectively evaluated with CEM, including acquisition of low-energy (LE) images and reconstructed images (RI) showing enhancement, concurrently with breast ultrasound (US) evaluation.
  Interventions: Diagnostic Test: Contrast-Enhanced Mammography
- retrospective cohort: The retrospective cohort will select the mammography and breast US data (BI-RADS score) of female patients with suspected breast abnormalities who had previous baseline matching.

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Mammography — Only patients in the prospective cohort will undergo CEM in addition to breast ultrasound.
  Groups: prospective cohort

SUMMARY:
Contrast-Enhanced Mammography (CEM) is a functional breast imaging technology. Like magnetic resonance imaging (MRI), CEM neovascularization enhancement can improve cancer detection rates, while lack of enhancement may lead to benign determination. The advantages of CEM are dramatically apparent in women with dense breasts. The purpose of this study was to investigate the additional diagnostic value of CEM added to the standard practice of mammography plus ultrasonography(US) in patients with suspicious breast lesions.

This study was a single-center prospective-retrospective combined observational study. In the prospective part, women with suspected breast abnormalities undergo prospective CEM evaluation, including acquisition of low energy (LE) images and recombined images (RI) showing enhancement, concurrently with breast US. The retrospective part selected the mammography and breast US data of female patients with suspected breast abnormalities who had previous baseline matching.

ELIGIBILITY:
Inclusion Criteria:

* Breast ultrasound or/and general mammography suggest that the lesion is BI-RADS 4 or above;
* Willing to undergo enhanced mammography examination;
* Agree to perform tumor core needle biopsy or excisional biopsy to confirm pathological diagnosis when necessary.

Exclusion Criteria:

* Allergy to iodinated contrast;
* Pregnant and lactating women;
* Suffering from kidney disease or abnormal kidney function, or undergoing renal dialysis;
* The breast is too large to be completely included in the full-field mammography examination at one time; ○5 Those with breast implants.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast lesions BI-RADS 4 and above treated at the Breast Surgery Department of Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
lesion biopsy rate | 2 years
  Total biopsy rate (including core needle biopsy and lesion excision biopsy) in patients with BI-RADS 4 and above with and without CEM.
breast cancer detection rate | 2 years
  Proportion of breast cancer detected among all patients undergoing biopsy.

SECONDARY OUTCOMES:
number of BI-RADS score upgrade | 3 years
  number of BI-RADS score upgrade during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yanna Zhang, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Department of Breast Surgery,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No